CLINICAL TRIAL: NCT00708292
Title: An Open-label, Multi-center, Phase I-Ib/II Study of AUY922 Administered as Single Agent and in Combination With Bortezomib With or Without Dexamethasone in Adult Patients in Relapse or Refractory Multiple Myeloma.
Brief Title: A Phase I-Ib/II Study to Determine the Maximum Tolerated Dose (MTD) of AUY922 Alone and in Combination With Bortezomib, With or Without Dexamethasone, in Patients With Relapsed or Refractory Multiple Myeloma.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAUY922A2103; 2007-006279-35 (EudraCT Number)
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2015-06

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: AUY922; Multiple Myeloma; HSP90 inhibitors; Phase I/II
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide; Bortezomib; Dexamethasone

ARMS (3):
- Single Agent AUY922 (Experimental)
  Interventions: Drug: AUY922
- AUY922 + Bortezomib (Experimental)
  Interventions: Drug: AUY922; Drug: Bortezomib
- AUY922 + Bortezomib + Dexamethasone (Experimental)
  Interventions: Drug: AUY922; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: AUY922
Drug: Bortezomib
  Arms: AUY922 + Bortezomib; AUY922 + Bortezomib + Dexamethasone
Drug: Dexamethasone
  Arms: AUY922 + Bortezomib + Dexamethasone

SUMMARY:
This is a Phase I-Ib/II, open-label, multicenter study of AUY922 administered intravenously in patients with multiple myeloma to determine the maximum tolerated dose. The Phase II part will investigate the efficacy of AUY922 in patients with multiple myeloma. Additionally, the study includes a Phase Ib combination part of AUY922 administered in combination with bortezomib, to determine the maximum tolerated dose of the combination drugs in patients with multiple myeloma.

ELIGIBILITY:
Inclusion criteria:

* Patients must have a diagnosis of active multiple myeloma.
* Phase I and Phase II part: Patients must have received at least 2 but not more than 4 prior line of therapy and their disease has progressed during or after last therapy.
* Phase Ib part: Patients must have received no more than 2 prior lines of therapy (excluding dexamethasone as single agent).
* ECOG Performance Status of ≤ 2.
* Patients must have acceptable neutrophil and platelet counts as well as adequate kidney and liver function.
* Patients must have magnesium levels above lower limit of normal or correctable with supplements.
* Patients must be willing and able to undergo bone marrow biopsy/aspirate.
* Able to sign informed consent.

Exclusion criteria:

* Prior treatment with any HSP90 or HDAC inhibitor for the treatment of multiple myeloma.
* Patients with unresolved diarrhea ≥ CTCAE grade 2.
* Patients with acute or chronic liver disease.
* Patients using medications that have a relative risk of prolonging the QT interval.
* Clinically significant cardiac diseases.
* Patients with known disorders due to a deficiency in bilirubin glucuronidation (e.g. Gilbert's syndrome).
* Pregnant or lactating women.
* Fertile women of childbearing potential (WCBP) not using adequate contraception.
* Male patients whose partners are WCBP, not using adequate contraception.
* Patients who unwilling or unable to comply with the protocol.
* Phase Ib part: Peripheral neuropathy ≥ CTCAE grade 1.
* Phase Ib part: Prior treatment with bortezomib.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2008-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The safe dose of AUY922 when administered once a week. | 54 weeks (Maximum Tolerated Dose (MTD))

SECONDARY OUTCOMES:
The safe dose of AUY922 when administered once a week in combination with bortezomib and dexamethasone. | 24 weeks (MTD determination of dual and triple combination)
Efficacy of AUY922 administered once a week alone and in combination | at baseline and every 2 cycles (time to document tumor progression)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (2):
  - Mayo Clinic - Arizona Cancer Clinical Research Unit, Scottsdale, Arizona
  - Cancer Therapy & Research Center / UT Health Science Center InstituteForDrugDevelopment(3), San Antonio, Texas
- Novartis Investigative Site, Melbourne, Australia
- Germany (3):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid

REFERENCES:
- [Derived] Seggewiss-Bernhardt R, Bargou RC, Goh YT, Stewart AK, Spencer A, Alegre A, Blade J, Ottmann OG, Fernandez-Ibarra C, Lu H, Pain S, Akimov M, Iyer SP. Phase 1/1B trial of the heat shock protein 90 inhibitor NVP-AUY922 as monotherapy or in combination with bortezomib in patients with relapsed or refractory multiple myeloma. Cancer. 2015 Jul 1;121(13):2185-92. doi: 10.1002/cncr.29339. Epub 2015 Mar 24. PMID 25809731
- See also: Results for CAUY922A2103 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6904